CLINICAL TRIAL: NCT01558947
Title: Peri-operative Chemotherapy With ECX (Epirubicin + Cisplatin + Capecitabine) or XP (Capecitabine + Cisplatin) in the Treatment of Advanced Gastric Cancer: a Randomized, Multicenter, Parallel Control
Brief Title: Peri-operative Chemotherapy With ECX or XP in the Treatment of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC-AGC-01
Record Dates: First submitted 2012-03-07; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; Peri-operative chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy with ECX (Experimental): chemotherapy with ECX
  Interventions: Drug: Peri-operative chemotherapy of ECX
- chemotherapy with XP (Experimental): chemotherapy with XP
  Interventions: Drug: Peri-operative chemotherapy of XP

INTERVENTIONS:
Drug: Peri-operative chemotherapy of ECX — Preoperative chemotherapy of ECX for 3 cycles(Epirubicin 50mg/m2 on day 1; capecitabine 1000mg/m2, 2 times / day, 1 to 14 days; cisplatin 60mg/m2 on day 1, need hydration, 21 day/cycle), operation after 2~4 weeks, and postoperative chemotherapy of ECX for 3 cycles 4~6 weeks after surgery.
  Other Names: ECX chemotherapy
  Arms: chemotherapy with ECX
Drug: Peri-operative chemotherapy of XP — Preoperative chemotherapy of XP for 3 cycles(capecitabine 1000mg/m2, 2 times / day, 1 to 14 days; cisplatin 60mg/m2 on day 1, need hydration, 21 day/cycle), operation after 2~4 weeks, and postoperative chemotherapy of XP for 3 cycles 4~6 weeks after surgery.
  Other Names: XP chemotherapy
  Arms: chemotherapy with XP

SUMMARY:
The purpose of this study is to evaluate the safety and the effect of perioperative chemotherapy in the treatment of advanced gastric cancer.

DETAILED DESCRIPTION:
To evaluate the security and the relapse-free survival time/rate(1,2,3 yrs) of perioperative chemotherapy with ECX (epirubicin + cisplatin + capecitabine) and XP (capecitabine + cisplatin）in advanced gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 to 70 years old.
* The preoperative evaluation: gastric cancer patients, ≥ T2 or N +; or staging II, IIIA, IIIB.
* Karnofsky score ≥ 70, life expectancy > 6 months.
* Endoscopic biopsy diagnosis of gastric cancer, excluding non-Hodgkin's lymphoma, leiomyosarcoma and other mesenchymal tumors.
* the blood and biochemical indicators of the subjects must meet the following criteria: Hb ≥ 9 g / dl; WBC ≥ 4,000 / mm3, ≤ 12000 / mm3; PLT ≥ 100,000/mm3; GOT, GPT within twice the institutional limit,serum total bilirubin < 1.5 times the upper limit of normal, serum creatinine< 1.25 times the upper limit of normal and creatinine clearance rate ≥ 60ml/min, LVEF ≥ 60%.
* have not received prior chemotherapy, radiotherapy and biological therapy.
* signed informed consent.
* must accept the standard D2 or D2 + radical gastrectomy.
* with good compliance.

Exclusion Criteria:

* pregnancy, breast-feeding women.
* allergy with chemotherapy drugs or metabolic disorder.
* the history of organ transplants (including bone marrow transplantation and autologous peripheral stem cell transplantation).
* had long received systemic steroid treatment (Note: short-term users of withdrawal > 2 weeks can be selected.)
* The existence of the peripheral nervous system disorders or significant neurological disorders and a history of central nervous system disorders.
* patients with severe infection requires treatment.
* patients associated with dysphagia, active peptic ulcer, incompleteness intestinal obstruction, active gastrointestinal bleeding, perforation.
* severe liver disease (such as cirrhosis), kidney disease, respiratory disease or uncontrollable diabetes.
* with other malignancies which were not cured.
* EKG abnormalities or heart disease with apparent clinical symptoms, including congestive heart failure, coronary heart disease with symptoms, uncontrollable arrhythmia, hypertension, and heart attack within 12 months or III or IV grade myocardial infarction. Coronary heart disease with symptoms, uncontrollable arrhythmia, hypertension, and heart attack within 12 months or III or IV grade myocardial infarction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
the relapse-free survival time/rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: xiangdong Cheng, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China